CLINICAL TRIAL: NCT06787261
Title: Involvement of Archaea in Carious Disease
Acronym: CARIARCHAE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RCAPHM24-0329
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Dental Caries
Keywords: Dental caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low risk of carriages (Experimental)
  Interventions: Other: saliva sample
- high risk for caries. (Other)
  Interventions: Other: saliva sample; Other: carious tissue samples

INTERVENTIONS:
Other: saliva sample — saliva sample
Other: carious tissue samples — carious tissue samples
  Arms: high risk for caries.

SUMMARY:
Dental caries is a major public health probleme the result of hard tissue demineralization and oral microbiota changes.

Methanogenic archaea, mainly Methanobrevibacter oralis, are associated with various oral problems, including pathologies periodontal.

Previous research has not really studied the Archaea in carious lesions, hence the importance of our study.

Our study aims to explore their potential role in the the development of caries by analysing their prevalence and their quantification in relation to the carious risk individual. The aim is to improve understanding of the Cavity microbiology to advance management of this pathology in terms of prevention or of treatment.

Our team is particularly competent in the field of Archaea, especially in the cultivation of Archaea methanogens since we have a dedicated platform. We also discovered the first human Nanoarchaea, opening up a whole new possible search field.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of legal age.
* Patient who is a beneficiary or entitled beneficiary of a social security
* Patient under the care of the Restorative and Preventive Dentistry of the PROMOD - Timone Dentistry Unit.
* Patients capable of giving written consent.

Exclusion Criteria:

Patient in a period of exclusion from another research protocol at the time of signing the consent form, Subjects covered by articles L1121-5 to 1121-8 of the Public Health public health code (minor patients, patients of full age under guardianship, patients deprived of their liberty, pregnant or breast-feeding), A person who does not have a sufficient command of reading and understanding of the French language to be able to consent to take part in the research Presence of periodontitis (gingivitis not being a criterion for a criterion for non-inclusion). Antibiotics taken in the previous month. Use of mouthwash in the previous 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Presence/absence of Archaea in participants' saliva samples. | 36 months

SECONDARY OUTCOMES:
Quantity of Archaea in the salivary sample of the participants. | 36 months
Viability/non-viability of Archaea in carious lesions | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: jean-olivier ARNAUD GENERAL DIRECTOR, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Asssistance Publique Hopitaux de Marseille, Marseille, France